CLINICAL TRIAL: NCT01664741
Title: Nicotine Dependence, Withdrawal and Replacement Therapy Assessed by PET Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00036996; R01DA026823 (NIH)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Nicotine Dependence
Keywords: Nicotine dependence; cigarette; smoking; nicotine replacement therapy; positron emission tomography
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nicotine patch - transdermal (Active Comparator): 21 mg nicotine patch
  Interventions: Drug: Nicotine patch - transdermal
- Placebo NRT (Placebo Comparator): Matching placebo patch
  Interventions: Drug: placebo
- Healthy non-smoker comparison (No Intervention): Demographically-matched women and men who have never smoked

INTERVENTIONS:
Drug: Nicotine patch - transdermal — 21 mg patch
  Other Names: Nicotine Replacement Therapy (NRT)
  Arms: Nicotine patch - transdermal
Drug: placebo
  Arms: Placebo NRT

SUMMARY:
The proposed research will provide significant new gender-specific information of scientific and clinical relevance on the function of the mu-opioid system in nicotine dependence and therapeutic effectiveness of nicotine replacement therapy (NRT). The studies will help to explain the differences in the prevalence of smoking in men and women, sex-specific differences in nicotine craving and withdrawal as well as the poorer therapeutic response to NRT. This work may pave the way to the design of improved pharmacotherapies that can more effectively target the endogenous opioid system in the treatment of nicotine dependence.

DETAILED DESCRIPTION:
While smoking prevalence has declined for both men and women over the last two decades, rates among women have shown a much shallower decrease and, in recent years, prevalence of cigarette initiation has been higher for girls than boys. Smoking among women of child-bearing age has significant negative health consequences for mother and child, increasing fetal and infant morbidity and mortality. Women are both less likely to initiate a quit attempt and more likely to relapse if these women do quit. Nicotine replacement therapy (NRT), still the most widely used smoking treatment intervention in the United States, is less effective for women compared with men, and women report less craving reduction on NRT. The endogenous opioid system is involved in smoking initiation, nicotine craving and reward as well as nicotine withdrawal symptoms. Interestingly, research suggests that sexual dimorphic features of the endogenous mu-opioid system may in part explain gender differences in nicotine effects. To better understand the role of the mu-opioid system in poorer NRT responses in women, this proposal will examine NRT effects on mu opioid receptor binding potential (MOR BP) in female compared to male smokers during active versus placebo NRT. Specifically, nicotine dependent women and men in active smoking status will undergo PET imaging for MOR BP measurement using 11C-carfentanil. Following baseline PET measurement in active smoking (scan 1), smokers will be randomized to active or placebo nicotine replacement therapy ((A-NRT or P-NRT); 72 hours later, a second scan will be obtained. As a reference group, demographically-matched women and men who have never smoked will undergo two scans as well. Behavioral measurements of nicotine reward, craving and withdrawal will be obtained repeatedly across the protocol. The proposed research will provide significant new, gender-specific information of scientific and clinical relevance on the function of the mu-opioid system in nicotine dependence and therapeutic effectiveness of nicotine replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* 21 - 60 years old
* must meet DSM-IV criteria for nicotine dependence and be actively smoking

Exclusion Criteria: subjects must meet study guidelines for medical and mental health status.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E McCaul, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 102 of the participants who passed the on-phone screen came in and signed the consent form to be enrolled in the study. Baseline characteristics data was collected from them but they however failed an assessment done prior to getting the PET scan and so could not start the study.
Groups:
- Nicotine Patch - Transdermal: 21 mg nicotine patch
  Nicotine patch - transdermal
- Placebo NRT: Matching placebo patch
  placebo
Period: Overall Study
Arm/Group | Nicotine Patch - Transdermal | Placebo NRT | Healthy Non-smoker Comparison
Started | 6 | 6 | 13
Completed | 6 | 6 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 102 of the participants who passed the on-phone screen came in and signed the consent form to be enrolled in the study. Baseline characteristics data was collected from them but they however failed an assessment done prior to getting the PET scan and so could not start the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Patch - Transdermal | Placebo NRT | Healthy Non-smoker Comparison | Total
Number analyzed (Participants) | 42 | 42 | 43 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 42 | 43 | 127
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 18 | 48
  Male | 27 | 27 | 25 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 6
  Not Hispanic or Latino | 37 | 38 | 42 | 117
  Unknown or Not Reported | 2 | 2 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 17 | 18 | 52
  White | 24 | 24 | 25 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 42 | 43 | 127
Years of regular smoking [Mean (Standard Deviation); unit: years] | 22.2 (12.8) | 22.2 (12.8) | 0 (0) | 22.2 (12.8)
Cigarettes per day [Mean (Standard Deviation); unit: number of cigarettes/day] | 17.0 (6.9) | 17.0 (6.9) | 0 (0) | 17.0 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mu-opioid Receptor Binding Potential (BP) Between Baseline and Post-patch Scans
Description: BP provides an estimate of the product of the density of available receptors (Bmax' or the receptor density Bmax less those occupied by endogenous transmitters) and the affinity [1/equilibrium dissociation constant (KD)]. We use reference tissue graphical analysis (RTGA) to obtain regional BP values using occipital lobe as a reference region. Negative BP change means means a decrease in the BP and positive BP change means an increase in the BP.
Time Frame: 90 minutes
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Nicotine Patch - Transdermal | Placebo NRT | Healthy Non-smoker Comparison
Number analyzed (Participants) | 6 | 6 | 13
ratio
  BP Change - Left Amygdala | -2.47 (3.91) | -5.94 (3.91) | 5.60 (2.66)
  BP Change - Ventral Striatum | -1.24 (3.50) | -9.25 (3.50) | 0.59 (2.38)

2. Secondary Outcome: Relationship Between Change in Mu-opioid Receptor Binding Potential and Visual Analog Craving Scale Score
Description: Regression measure (β) between change in mu-opioid receptor binding potential between baseline scan and post-treatment scan in the left amygdala and mean Craving Visual Analog Scale score on Days 2 - 4 of the Clinical Research Unit stay. Craving visual analog scale ranges from 0 (not at all) to 20 (worst ever).
Time Frame: 72 hours
Population: This assessment was not done on the healthy non-smokers because they didn't have any nicotine craving.
Measure: Number; unit: unitless
Arm/Group | Nicotine Patch - Transdermal | Placebo NRT | Healthy Non-smoker Comparison
Number analyzed (Participants) | 6 | 6 | 0
unitless | 0.556 | -0.550 |

3. Secondary Outcome: Relationship Between Change in Mu-opioid Receptor Binding Potential and Minnesota Nicotine Withdrawal Scale Score
Description: Regression measure (β) between change in mu-opioid receptor binding potential between baseline scan and post-treatment scan and mean Minnesota Nicotine Withdrawal Scale (MNWS) score on Days 2 - 4 of the Clinical Research Unit stay. The MNWS is a self-report measure that consists of 14 nicotine withdrawal symptoms each rated on a 0 - 4 response scale for severity over the past 24 hours. Higher scores are indicative of greater nicotine withdrawal severity.
Time Frame: 72 hours
Population: This assessment was not done on the healthy non-smokers because they didn't have any nicotine craving.
Measure: Number; unit: unitless
Arm/Group | Nicotine Patch - Transdermal | Placebo NRT | Healthy Non-smoker Comparison
Number analyzed (Participants) | 6 | 6 | 0
unitless
  Left Amygdala | -0.087 | -0.836 |
  Ventral Striatum | 0.419 | -0.794 |

ADVERSE EVENTS:
Time Frame: During 4 day Clinical Research Unit stay
Arm/Group | Nicotine Patch - Transdermal | Placebo NRT
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT01664741/Prot_SAP_000.pdf